CLINICAL TRIAL: NCT01666301
Title: Reticulocyte Dynamic and Related Hemoglobin Variability in Hemodialysis Patients Treated With Darbepoetin Alfa and C.E.R.A.: a Randomized Controlled Trial
Brief Title: ESAs, Reticulocyte Dynamic and Hemoglobin Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Regionale di Locarno (Other)
Responsible Party: Principal Investigator, Luca Gabutti, MD, Head of Department; internal medicine, Ospedale Regionale di Locarno
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Epo-Loc1
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Erythropoiesis Stimulating Agent Pharmacodynamics
Keywords: Erythropoietin stimulating agents; Hemoglobin; Reticulocytes; Variability

ARMS (2):
- C.E.R.A. (Active Comparator): C.E.R.A. every 4 and then every 2 weeks
  Interventions: Drug: comparison between darbepoetin alfa and C.E.R.A. and different administration intervals
- Darbepoetin (Active Comparator): Darbepoetin alfa every 4 and then every 2 weeks
  Interventions: Drug: comparison between darbepoetin alfa and C.E.R.A. and different administration intervals

INTERVENTIONS:
Drug: comparison between darbepoetin alfa and C.E.R.A. and different administration intervals

SUMMARY:
Background: In a simulation based on a pharmacokinetic model we demonstrated that increasing the erythropoiesis stimulating agents (ESAs) half-life or shortening their administration interval decreases hemoglobin variability. The benefit of reducing the administration interval was however lessened by the variability induced by more frequent dosage adjustments. The purpose of this study was to analyze the reticulocyte and hemoglobin kinetics under different ESAs and administration intervals in a collective of chronic hemodialysis patients.

Methods: The study was designed as an open-label, randomized, four-period cross-over investigation, including 30 patients under chronic hemodialysis at the regional hospital of Locarno (Switzerland) in September 2009 and lasting 2 years. Four treatment strategies (C.E.R.A. every 4 weeks Q4W and every 2 weeks Q2W, Darbepoetin alfa Q4W and Q2W) were compared with each other. The mean square successive difference of hemoglobin, reticulocyte count and ESAs dose was used to quantify variability. We distinguished a short- and a long-term variability based respectively on the weekly and monthly successive difference.

ELIGIBILITY:
Inclusion Criteria:

* chronic patients aged 18 years or older, undergoing dialysis 3 times a week for at least 8 weeks before screening, necessitating continuous subcutaneous treatment with weekly Darbepoetin alfa or Erythropoietin beta to maintain hemoglobin (Hb) targets

Exclusion Criteria:

* pregnancy; not respecting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
hemoglobin variability | 2 years

SECONDARY OUTCOMES:
differences in reticulocyte count over time | 2 years
risk of hemoglobin overshooting (HR) | 2 years
superiority of every 2 week administration | 2 years
reticulocyte variability | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gabutti, MD, Principal Investigator — Ospedale Regionale Locarno
Locations (1):
- Ospedale Regionale Locarno, Locarno, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Forni V, Bianchi G, Ogna A, Salvade I, Vuistiner P, Burnier M, Gabutti L. Reticulocyte dynamic and hemoglobin variability in hemodialysis patients treated with Darbepoetin alfa and C.E.R.A.: a randomized controlled trial. BMC Nephrol. 2013 Jul 22;14:157. doi: 10.1186/1471-2369-14-157. PMID 23870287